CLINICAL TRIAL: NCT02009722
Title: Intrathecal Opioids for Pain Control After Cesarean Delivery: Determining the Optimal Dose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hans P. Sviggum, M.D., Assistant Professor of Anesthesiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-008490
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Analgesia, Obstetrical; Cesarean Section
Keywords: Cesarean Delivery; Intrathecal Morphine; Intrathecal Hydromorphone; Obstetrical Analgesia; Spinal Anesthesia
MeSH Terms: conditions — Agnosia | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal hydromorphone (Active Comparator): Patients will be randomized to receive a one-time dose of intrathecal hydromorphone or intrathecal morphine as part of their spinal anesthesia. The starting dose of intrathecal hydromorphone will be 40 micrograms. This will be adjusted in subsequent patients based on the previous patient's success or failure according to an up-and-down methodology utilizing a biased coin design.
  Interventions: Drug: Hydromorphone
- Intrathecal morphine (Active Comparator): Patients will be randomized to receive a one-time dose of intrathecal hydromorphone or intrathecal morphine as part of their spinal anesthesia. The starting dose of intrathecal morphine will be 100 micrograms. This will be adjusted in subsequent patients based on the previous patient's success or failure according to an up-and-down methodology utilizing a biased coin design.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Duramorph is administered as part of spinal anesthesia for post-operative pain relief.
  Other Names: Duramorph
  Arms: Intrathecal morphine
Drug: Hydromorphone — Hydromorphone (Dilaudid) is administered in the intrathecal space for post-operative pain control
  Other Names: Dilaudid
  Arms: Intrathecal hydromorphone

SUMMARY:
Both hydromorphone and morphine are administered as part of spinal anesthesia to help improve pain control after cesarean delivery. In this study, the investigators are going to determine the doses of each of those medicines that provides optimal pain control to women undergoing cesarean delivery while limiting side effects related to those medicines. The investigators hypothesize that the doses of hydromorphone and morphine that provide optimal pain control without significant side effects will be 100 micrograms and 150 micrograms, respectively. The investigators further hypothesize that at each respective optimal dose, side effects will be less in the hydromorphone group.

DETAILED DESCRIPTION:
Spinal anesthesia is the most common anesthetic technique used for Cesarean delivery in the United States and across the world. Intrathecal opioids are administered along with a local anesthetic during spinal anesthesia for Cesarean delivery to provide postoperative analgesia. The effectiveness of intrathecal morphine for post-Cesarean pain control is well established, but the effectiveness of intrathecal hydromorphone in this patient population is limited to case reports and small retrospective studies. No prospective studies have been conducted to establish the effectiveness of intrathecal hydromorphone for post-Cesarean pain.

Hydromorphone has been studied extensively as a substitute for intrathecal morphine in patients with chronic noncancer pain. In fact, a recent consensus article placed hydromorphone as a first line therapy along with morphine for intrathecal pain management. Its ability to treat post-Cesarean pain when administered in the epidural space has been known for quite some time, but its effects in the intrathecal space are less established. In patients undergoing Cesarean delivery, intrathecal doses of 40 to 100 micrograms have been reported to provide good pain scores postoperatively with only minimal side effects. Doses of up to 300 micrograms have been used, leading to excellent pain control without out respiratory depression, but with significant pruritus and nausea.

Although reducing pain, intrathecal opioids are associated with side effects including pruritus, nausea, and respiratory depression. A meta-analysis reviewing twenty-eight studies which investigated intrathecal morphine versus placebo demonstrated moderate increases in the incidences of pruritus, nausea and vomiting. In fact the incidence of nausea with IT morphine has been reported to be 33%. While hydromorphone is similar chemically to morphine, it is metabolized differently. Differences in pharmacokinetics may allow for differences in side effect profiles. Hydromorphone is more lipid soluble than morphine. This decreases its spread within the intrathecal space and enhances its penetration into the dorsal horn of the spinal cord where interactions with opioid receptors occur. Some studies have found that hydromorphone causes less nausea and pruritus than morphine, while others have not. Although opioid-induced respiratory depression is a rare event, studies evaluating intrathecal hydromorphone for post-Cesarean delivery pain have not reported any cases of respiratory depression.

The optimal dose of intrathecal morphine for analgesia following Cesarean delivery is still debated and the efficacy of intrathecal hydromorphone has not been studied extensively in this patient population. The investigators aim to identify the dose of each medication that provides good pain relief without causing significant side effects. The investigators will then perform a comparative analysis of each drug at their optimal dose.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting for elective cesarean delivery with no major co-morbidities, including pregnancy induced co-morbidities (e.g. pre-eclampsia)
* Singleton gestation at term (37-42 weeks)
* Desire to have a spinal anesthesia technique for cesarean delivery

Exclusion Criteria:

* Current or historical evidence of clinically significant medical disease or condition
* Any contraindication to the administration of a spinal technique for anesthesia
* History of hypersensitivity or idiosyncratic reaction to opioid medications
* Chronic pain syndrome or current regular opioid use
* Evidence of anticipated fetal anomalies
* Allergy or intolerance to Tylenol, ketorolac, ibuprofen, or oxycodone
* BMI > 40

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans P Sviggum, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Rochester Methodist Hospital, Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Beatty NC, Arendt KW, Niesen AD, Wittwer ED, Jacob AK. Analgesia after Cesarean delivery: a retrospective comparison of intrathecal hydromorphone and morphine. J Clin Anesth. 2013 Aug;25(5):379-383. doi: 10.1016/j.jclinane.2013.01.014. Epub 2013 Aug 17. PMID 23965210
- [Background] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Background] Rauch E. Intrathecal hydromorphone for postoperative analgesia after cesarean delivery: a retrospective study. AANA J. 2012 Aug;80(4 Suppl):S25-32. PMID 23248827
- [Background] Rauch E. Intrathecal hydromorphone for cesarean delivery: in search of improved postoperative pain management: a case report. AANA J. 2011 Oct;79(5):427-32. PMID 23256273
- [Background] Terajima K, Onodera H, Kobayashi M, Yamanaka H, Ohno T, Konuma S, Ogawa R. Efficacy of intrathecal morphine for analgesia following elective cesarean section: comparison with previous delivery. J Nippon Med Sch. 2003 Aug;70(4):327-33. doi: 10.1272/jnms.70.327. PMID 12928713
- [Background] Gehling M, Tryba M. Risks and side-effects of intrathecal morphine combined with spinal anaesthesia: a meta-analysis. Anaesthesia. 2009 Jun;64(6):643-51. doi: 10.1111/j.1365-2044.2008.05817.x. PMID 19462494
- [Background] Dougherty TB, Baysinger CL, Henenberger JC, Gooding DJ. Epidural hydromorphone with and without epinephrine for post-operative analgesia after cesarean delivery. Anesth Analg. 1989 Mar;68(3):318-22. PMID 2465709
- [Background] Pace NL, Stylianou MP. Advances in and limitations of up-and-down methodology: a precis of clinical use, study design, and dose estimation in anesthesia research. Anesthesiology. 2007 Jul;107(1):144-52. doi: 10.1097/01.anes.0000267514.42592.2a. PMID 17585226
- [Background] Gerancher JC, Floyd H, Eisenach J. Determination of an effective dose of intrathecal morphine for pain relief after cesarean delivery. Anesth Analg. 1999 Feb;88(2):346-51. doi: 10.1097/00000539-199902000-00023. PMID 9972754

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Started | 41 | 43
Received Intervention | 41 | 42
Completed | 40 | 40
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Did not receive intervention | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (4.1) | 30.6 (4.3) | 30.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose of IT Morphine and IT Hydromorphone for Adequate Analgesia (Pain Score Less Than or Equal to 3) in 90% of Patients
Description: Each patient will be interviewed by a member of the study team 12 hours after receiving their spinal anesthetic (which will include either hydromorphone or morphine). Patients will be asked to rate their current level of pain on a scale of 0 (no pain) to 10 (worst pain imaginable). A pain score <4 will be considered a success. The up-down sequential allocation method will be used to determine the dose (mcg) of IT hydromorphone and IT morphine for subsequent patients
Time Frame: 12 hours after administration of spinal anesthesia
Population: The primary outcome was determining the optimal dose of IT morphine and IT hydromorphone for patients undergoing cesarean delivery. Study was designed to determine the ED90 (effective dose in 90% patients; effective dose meaning a VAS score for pain of 3 or less at 12 hours after spinal placement).
Measure: Number; unit: micrograms
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 40 | 40
micrograms | 75 | 150

2. Secondary Outcome: Side Effects: Pruritus
Description: Patients will be evaluated by a member of the study team at 6 hours after spinal administration. The number of patients with moderate or severe pruritus will be recorded.
Time Frame: 6 hours after spinal administration
Population: The number of patients at the most commonly used doses of IT medication (50, 75, 100 mcg for hydromorphone) and (100, 150 mcg) for morphine were used in analysis
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 33 | 39
participants | 23 | 19

3. Secondary Outcome: Side Effects: Nausea
Description: Patients will be evaluated by a member of the study team at 6 hours after spinal administration. Patients with moderate or severe nausea will be recorded.
Time Frame: 6 hours after spinal
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 33 | 39
participants | 11 | 16

4. Secondary Outcome: Side Effects: Sedation
Description: Patients will be evaluated by a member of the study team at 6, 12, and 24 hours after spinal administration. The presence of sedation will be graded by the Richmond Agitation Sedation Scale. Patients with a score of (-)2 or lower on the Richmond were classified as being positive for sedation.
Time Frame: 6, 12, and 24 hours after spinal administration
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 40 | 40
participants | 0 | 0

5. Secondary Outcome: Pruritus
Description: Patients will be evaluated by a member of the study team at 12 hours after spinal administration. The number of patients with moderate or severe pruritus will be recorded.
Time Frame: 12 hours after spinal
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 33 | 39
participants | 10 | 9

6. Secondary Outcome: Pruritus
Description: Patients will be evaluated by a member of the study team at 24 hours after spinal administration. The number of patients with moderate or severe pruritus will be recorded.
Time Frame: 24 hours after spinal
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 33 | 39
participants | 8 | 8

7. Secondary Outcome: Nausea
Description: Patients will be evaluated by a member of the study team at 12 hours after spinal administration. The number of patients with moderate or severe nausea will be recorded.
Time Frame: 12 hours after spinal
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 33 | 39
participants | 7 | 5

8. Secondary Outcome: Nausea
Description: Patients will be evaluated by a member of the study team at 24 hours after spinal administration. The number of patients with moderate or severe nausea will be recorded.
Time Frame: 24 hours after spinal
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 33 | 39
participants | 1 | 4

9. Secondary Outcome: Treatment for Nausea
Description: number of patients needing medication treatment for nausea in first 24 hours
Time Frame: First 24 hours
Population: patients receiving most commonly used doses of IT medication (50,75,100 mcg for hydromorphone; 100, 150 mcg for morphine)
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 33 | 39
participants | 13 | 17

10. Secondary Outcome: Treatment for Pruritus
Description: The number of patients needing medical treatment for pruritus in first 24 hours after surgery
Time Frame: First 24 hours after spinal
Population: only patients receiving most commonly used doses of IT hydromorphone (50,75,100 mcg) and morphine (100,150 mcg)
Measure: Number; unit: participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 33 | 39
participants | 8 | 4

ADVERSE EVENTS:
Description: Hydromorphone arm: 41 patients received the intervention, 40 were analyzed
  Morphine arm: 43 patients were randomized to this arm, 42 received the intervention (thus the denominator for adverse events) and 40 were analyzed
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 29/41 | 26/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrathecal Hydromorphone (N=41) | Intrathecal Morphine (N=42)
Moderate to Severe Pruritus (Skin and subcutaneous tissue disorders) | 27 (27) | 22 (22) — Patients experiencing moderate to severe pruritus (self-reported) within 24 hours of spinal administration
Moderate to Severe Nausea (Gastrointestinal disorders) | 13 (13) | 17 (17) — Patients experiencing moderate to severe nausea (self-reported) within 24 hours of spinal administration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes